CLINICAL TRIAL: NCT00485212
Title: The Effect of a Compression Bandage in Local Infiltration Analgesia After Total Knee Arthroplasty
Brief Title: Compression Bandage in Local Infiltration Analgesia Afte Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF01327078
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-05

CONDITIONS: Total Knee Arthroplasty
Keywords: postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: compression bandage

SUMMARY:
purpose: to determine wether a compression bandage prolongs analgesia of local infiltration analgesia after total knee arthroplasty

DETAILED DESCRIPTION:
patients are randomised to receive a compression bandage or a non-compression bandage

ELIGIBILITY:
Inclusion Criteria:

* scheduled for total knee arthroplasty
* speak and understand Danish

Exclusion Criteria:

* severe obesity
* allergies to local anaesthetics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
pain, Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Andersen, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark